CLINICAL TRIAL: NCT00572637
Title: An Open-Label, Dose-escalation, Phase I Study to Determine the Maximum Tolerated Dose, Recommended Dose, Pharmacokinetics, and Pharmacodynamics of the Proteosome Inhibitor CEP 18770 Given Intravenously as Single Agent in Patients With Advanced Solid Tumours or Non-Hodgkin's Lymphomas
Brief Title: Phase I Study of the Proteosome Inhibitor CEP 18770 in Patients With Solid Tumours or Non-Hodgkin's Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ethical Oncology Science (Industry)
Responsible Party: Gabriella Camboni, VP Development, EOS (Ethical Oncology Science)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-CEP\I\01
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-05

CONDITIONS: Solid Tumors; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — delanzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CEP-18770 — Administered as intravenous infusion on days 1, 4, 8, and 11 of a 21-day cycle up to 6 cycles. Starting dose 0,1 mg/sqm

SUMMARY:
This Phase 1 escalating-dose study is designed to assess, the safety, tolerability, pharmacokinetics, and pharmacodynamics of the novel proteasome inhibitor CEP 18770, given intravenously as single agent, in patients with advanced, incurable solid tumours or NHL, and to identify the recommended dose of CEP 18770 to be used in Phase 2 studies.

DETAILED DESCRIPTION:
This is an open-label, multicenter, dose-escalating study to determine the MTD and dose limiting toxicities (DLTs) of CEP 18770, a novel proteasome inhibitor. The study will also characterize the pharmacokinetics and the pharmacokinetic/pharmacodynamic relationship of CEP 18770, and assess the safety and tolerability of CEP-18770 treatment as well as any effect on tumour response whenever possible.

Patients will be treated intravenously with CEP 18770 on days 1, 4, 8, and 11 of a 21-day cycle period. Additional cycles may be administered, up to 6, as long as patients are maintaining their performance status and appear to be receiving clinical benefit from the study.

Safety data will be collected for all patients in order to determine the toxicity and reversibility of toxicity of CEP 18770. Formal assessments will be performed throughout the study including at baseline, prior to each dose of study medication every week, and 30 days following the last dose of study drug. Patients with drug-related toxicities will continue to be reviewed until resolution or stabilization of the toxicity. Pharmacokinetic and pharmacodynamic parameters will also be assessed in each cohort of patients during cycle 1. Where applicable, tumour measurements will be documented and any observed anti-tumour activity will be evaluated.

The study will follow a conventional MTD design with patients recruited in cohorts of 3 patients, with criteria to expand to 6 patients. Enrolment for each cohort will begin when the required number of patients in the prior cohort have completed one 21-day cycle of study drug treatment at the current dose level without experiencing a DLT. Once the MTD has been determined, additional 10 patients will be treated at the MTD to further explore the toxicity of this dose, and its suitability for Phase II studies.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of relapsed or refractory solid tumour or non-Hodgkin's lymphoma
* unresponsive or poorly responsive to accepted treatment modalities
* expected survival of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
* fully recovered from any prior surgical procedure(s) and from reversible side effects of prior therapy for cancer including radiation therapy, chemotherapy, and immunotherapy (exceptions: alopecia and grade 1 neurotoxicity).
* al least 4 weeks from last cancer therapy (or 6 weeks from previous mitomycin C; 2 weeks from previous biological therapy; 8 weeks from previous bevacizumab)
* no more than 3 previous chemotherapies for advanced disease (excluding TKIs)
* good health as determined by a medical and psychiatric history, medical examination, ECG, serum chemistry, hematology, urinalysis, and serology.
* for women of childbearing potential use of a medically accepted method of contraception for the duration of the study and for 60 days after the last administration of study drug
* for men not surgically sterile use of an accepted method of birth control for the duration of the study and for 60 days after the last administration of study drug
* willingness and ability to comply with study requirements

Exclusion Criteria:

* Any of the following hematologic values: absolute neutrophil count (ANC) less than 1500/mm3, platelet count less than 100,000/mm3, or hemoglobin less than 9 g/dL
* Any of the following hepatic function values: bilirubin greater than 1.5 times the upper limit of normal (ULN) or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 times the ULN
* Serum creatinine value greater than 1.5 mg/dL.
* Known cerebral metastases or active CNS disease
* Signs indicating potential major bone marrow involvement
* Significant neurotoxicity (higher than grade 1 as defined by NCI-CTC scale v. 3.0 and/or a TNSc value ≥ 3)
* Any concomitant cancer related treatment. (Continuing endocrine treatment at stable doses is allowed; treatment must be ongoing for at least 4 weeks)
* Concomitant treatment with steroids
* Previous treatment with high-dose chemotherapy with PBSC support
* Any investigational drug within the past 4 weeks
* Any medications which are human cytochrome P450 34A (CYP3A4) substrates within 1 week, or 5 half-lives (whichever is longer) before the first administration of study drug or need for continuous treatment with these medications during the study
* Known hypersensitivity to boronic acid derivatives or excipients in the CEP-18770 formulation.
* Any condition which, in the judgment of the Investigator, would place the subject at undue risk or interfere with the results of the study, or make the subject otherwise unsuitable (e.g., risk factors for neurological toxicities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) and Maximum Tolerated Dose (MTD) of CEP 18770 | Within the first 21-day cycle

SECONDARY OUTCOMES:
Pharmacokinetics of CEP-18770 following single and multiple dose administration. | Within the first 21-day cycle
Profile and time course of inhibition and recovery of proteasome activity | Within the first 21-day cycle
Antineoplastic activity evaluated with internationally accepted response criteria | throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Cristiana Sessa, MD, PhD, Principal Investigator — Oncology Institute of Southern Switzerland - Ospedale S. Giovanni Bellinzona CH
Locations (3):
- Europen Institute of Oncology, Milan, Italy
- Switzerland (2):
  - IOSI - Oncology Institute of Southern Switzerland - Ospedale S. Giovanni, Bellinzona
  - Kantonsspital St. Gallen, Sankt Gallen